CLINICAL TRIAL: NCT03039816
Title: A Nasally Applied Cellulose Powder in Seasonal Allergic Rhinitis in Adults With Grass Pollen Allergy: A Double-Blind, Randomised, Placebo-Controlled, Parallel-Group Study
Brief Title: Cellulose Powder Against Grass Pollen Allergic Rhinitis
Acronym: CPARGPDBPC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nasaleze International Ltd (Industry)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIL001/2013
Record Dates: First submitted 2016-12-12; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): The patients were randomly assigned to active (Nasaleze cellulose powder) or placebo groups using an identical device to be puffed in each nostril 3 times daily. The nasal powders were supplied in plastic containers, which deliver the powder from a nozzle when squeezed. The exact amount delivered is not standardized and the variation in the patterns of deposition in the nose is not known. The placebo was a lactose powder with the same particle size, appearance and the same tinge of mint taste as the cellulose powder.
  Interventions: Device: Nasaleze
- Placebo (Placebo Comparator): The patients were randomly assigned to active or placebo groups using an identical device to be puffed in each nostril 3 times daily. The nasal powders were supplied in plastic containers, which deliver the powder from a nozzle when squeezed. The exact amount delivered is not standardized and the variation in the patterns of deposition in the nose is not known. The placebo was a lactose powder with the same particle size, appearance and the same tinge of mint taste as the cellulose powder.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Nasaleze — Nasaleze cellulose powder
  Other Names: Nasaval
  Arms: Active
Device: Placebo — Lactose powder in the same plastic container as Nasaleze and with the same taste
  Arms: Placebo

SUMMARY:
Background: A nasally applied cellulose powder is increasingly used in many countries as a remedy for allergic rhinitis. In 2009, a 4-week study in birch pollen-allergic children showed a reduction in nasal symptoms. The best effect occurred on days with lower pollen counts. The present study in grass pollen-allergic adults used the same basic design. Methods: In May 2013, a double-blind, placebo-controlled study was conducted in 108 patients with allergic rhinitis due to grass pollen (18-40 years of age). SMS on mobile phones were used as reminders of treatment and reporting of symptom scores.

DETAILED DESCRIPTION:
The study was performed at university clinics in Kharkiv and Dnepropetrovsk in Ukraine in May 2013. 108 subjects 18-40 years of age were recruited locally to 2 centres. They all had a history of typical symptoms of seasonal allergic rhinitis (SAR) during late spring - early summer. At first appointment the history was scrutinized and an assessment of the severity excluded previous use of nasal steroids or a current need for nasal steroids. They should not have perennial symptoms or a history of asthma. They were tested with a blood sample for ImmunoCAP Specific Immunoglobulin E (IgE) for timothy grass pollen and birch pollen, with >0.35 Kilounits (kU)/ml counted as positive.

The patients were randomly assigned to active or placebo in groups using an identical device to be puffed in each nostril 3 times daily. The nasal powders were supplied in plastic containers, which deliver the powder from a nozzle when squeezed. The exact amount delivered is not standardized and the variations of patterns of deposition in the nose are not known. The placebo was a lactose powder with the same particle size, appearance and the same tinge of mint taste as the cellulose powder.

Rescue medication could be obtained by the investigators after emergency contacts. Oral antihistamine was loratadine 10 mg tablets and sodium chromoglycate eye drops. Each subject obtained oral and written instructions about the SMS. The SMS-reporting of symptoms started with a run in period for 3 days before the treatment and lasted for the 4 weeks of treatment during the grass pollen season

Three times a day the patients were reminded by SMS to take their nasal puffs and were asked to confirm the intake by a response SMS. In the evening, they were asked about the severity of symptoms during the preceding day from the nose, eyes and lower airways and to answer with a figure 1-6, corresponding to 1 "no trouble at all", 2"little trouble", 3"moderate trouble", 4"rather much trouble", 5"much trouble", and 6 "very much trouble" respectively. From the nose, scoring of sneezing, running nose and blocked nose were reported. For the eyes and lower airways, respectively, only a concluding figure was used.

In the registration a question was added daily on the use of rescue medication.

At a concluding appointment after the treatment period, the subjects were asked about their global opinion of the efficacy: No effect, good effect, very good effect. They also were asked whether they believed they had obtained the active substance or placebo.

The study was performed at university clinics in Kharkiv and Dnepropetrovsk in Ukraine in May 2013. 108 subjects 18-40 years of age were recruited locally to 2 centres. They all had a history of typical symptoms of SAR during late spring - early summer. At first appointment the history was scrutinized and an assessment of the severity excluded previous use of nasal steroids or a current need for nasal steroids. They should not have perennial symptoms or a history of asthma. They were tested with a blood sample for ImmunoCAP Specific IgE for timothy grass pollen and birch pollen, with >0.35 kU/ml counted as positive.

The patients were randomly assigned to active or placebo in groups using an identical device to be puffed in each nostril 3 times daily. The nasal powders were supplied in plastic containers, which deliver the powder from a nozzle when squeezed. The exact amount delivered is not standardized and the variations of patterns of deposition in the nose are not known. The placebo was a lactose powder with the same particle size, appearance and the same tinge of mint taste as the cellulose powder.

Rescue medication could be obtained by the investigators after emergency contacts. Oral antihistamine was loratadine 10 mg tablets and sodium cromoglycate eye drops. Each subject obtained oral and written instructions about the SMS. The SMS-reporting of symptoms started with a run in period for 3 days before the treatment and lasted for the 4 weeks of treatment during the grass pollen season

Three times a day the patients were reminded by SMS to take their nasal puffs and were asked to confirm the intake by a response SMS. In the evening, they were asked about the severity of symptoms during the preceding day from the nose, eyes and lower airways and to answer with a figure 1-6, corresponding to 1 "no trouble at all", 2"little trouble", 3"moderate trouble", 4"rather much trouble", 5"much trouble", and 6 "very much trouble" respectively. From the nose, scoring of sneezing, running nose and blocked nose were reported. For the eyes and lower airways, respectively, only a concluding figure was used.

In the registration a question was added daily on the use of rescue medication.

At a concluding appointment after the treatment period, the subjects were asked about their global opinion of the efficacy: No effect, good effect, very good effect. They also were asked whether they believed they had obtained the active substance or placebo.

Statistical methods For each question the mean score was calculated for the whole 28 days period for every subject. Mean values for the sum of all scores as well as the sum of the nasal scores were also calculated. The scores from the two treatment groups were then compared using t-tests. The group comparison of reflective opinions and the guess on obtained medication at the follow up visit were assessed using the Chi-square test.

The concluding opinion at the follow up visit were analysed using the chi-square test.

The study was approved by the local ethics committees at the respective hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a history of typical symptoms of hay fever during late spring or early summer
* Mild or moderate severity of symptoms of seasonal allergic rhinitis.
* Positive allergy test for grass pollen allergy.
* Voluntarily given written informed consent to study participation encompassing consent to data recording and verification procedures;
* Patients are able and willing to comply with the requirements of the study protocol.
* Patients who have not received any pollen disease treatment for one week prior to the study.

Exclusion Criteria:

* Previous treatment with nasal steroids or current indications for the administration of nasal steroids.
* Nasal symptoms during all seasons of the year or during spring time preceding the grass pollen season.
* Clinical signs of predominating nasal obstruction. The patient must be judged to be able to reach the nasal cavity with the study powder.
* Other respiratory or chronic diseases.
* Previous use of the study product
* Inability to give informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Symptoms of allergic rhinitis | Day 1-28 of treatment period
  Group total of symptoms scored retrospectively once daily

SECONDARY OUTCOMES:
Adverse events | Day 1-28 and day 32
  Answer on daily question on Short Message Service (SMS) during treatment and supplementing interview at concluding appointment
Use of rescue medication | Treatment period day 1-28
  Daily answer on SMS question on possible use of rescue medication
Global opinion of the efficacy | Day 32, after completed treatment
  Questions on alternatives "No effect, good effect, very good effect
Guess on obtained treatment | Day 32, after completed treatment
  Question on whether they believed they had obtained the active substance or placebo.

CONTACTS AND LOCATIONS:
Locations (3):
- Departments of Pediatrics and Biological and Environmental Sciences, Gothenburg, Sweden
- Ukraine (2):
  - Mechanikov Dnipropetrovsk Regional Clinical Hospital, Departmnet of Profpathology, Zhovteneva sq 14, Dnipro
  - Kharkiv National Medical University Department of Internal medicine propedeutics No 2 4 Lenin str, Kharkiv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aberg N, Ospanova ST, Nikitin NP, Emberlin J, Dahl A. A nasally applied cellulose powder in seasonal allergic rhinitis in adults with grass pollen allergy: a double-blind, randomized, placebo-controlled, parallel-group study. Int Arch Allergy Immunol. 2014;163(4):313-8. doi: 10.1159/000360734. Epub 2014 Apr 29. PMID 24852424